CLINICAL TRIAL: NCT06612762
Title: Effect of Naringenin Supplementation on the Speed of Bone Fusion and the Concentration of Plasma Inflammatory Factors in Patients With Bone Fractures.
Brief Title: Naringenin Supplementation in Bone Fracture Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Associate Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 43008307
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-11

CONDITIONS: Bone Fractures
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naringenin (Experimental): The daily ingestion of capsules containing naringenin
  Interventions: Dietary Supplement: The daily ingestion of capsules containing naringenin
- Control (Placebo Comparator): Patients will receive placebo capsules

INTERVENTIONS:
Dietary Supplement: The daily ingestion of capsules containing naringenin — Following surgical intervention, patients will be administered two capsules (equivalent to 500 mg) daily for a period of 14 days. Subsequently, patients will ingest the maintenance dose of 250 mg per day until the 90th day post-surgery.
  Arms: Naringenin
Dietary Supplement: Placebo — The daily ingestion of capsules containing placebo

SUMMARY:
Fractures of the lower extremities represent a significant proportion of injuries sustained by polytrauma patients, with a notable association with prolonged hospitalization, chronic disability, and impaired physical functioning. The occurrence of surgical site infections (SSI) represents a significant threat to the efficacy of osteosynthesis procedures. As with other traumas and surgical procedures, the secretion of inflammatory mediators is markedly elevated in this cohort of patients following surgery. Naringenin is one of the most prevalent flavonoids, occurring naturally in grapefruit and other citrus fruits. In vitro studies have demonstrated that naringenin may stimulate the release of osteogenic cytokines and suppress the production of pro-inflammatory factors, which can result in a reduction in bone resorption. Based on these findings, naringenin may prove an effective agent for accelerating the rate of fusion and controlling inflammation. Furthermore, it may enhance quality of life and augment functional activity.

DETAILED DESCRIPTION:
The study subjects will be selected from among the patients with bone fractures of the lower limbs who are hospitalized in the orthopedic department of Ayatollah Taleghani University Hospital in Tehran. The following criteria will be used to determine which patients are eligible for inclusion in the study:

Inclusion criteria: patients aged 18 to 60 years, candidates for orthopedic surgery for bone fractures of the lower limbs, ambulatory without assistance for a minimum of two months prior to the fracture, not having undergone amputation of the lower limbs, not suffering from liver cirrhosis, not suffering from advanced kidney failure (blood creatinine higher than 1.4 mg/dL), not having metastatic cancer. Additionally, subjects must not have any chronic inflammatory diseases, nor must they be taking any drugs that affect bone metabolism, including calcitonin, bisphosphonates, and corticosteroids. Furthermore, subjects must not be taking any anti-inflammatory drugs.

Subjects will be excluded from the study if they experience an allergic or intolerant reaction to Narangenin capsules, if there are any abnormal changes in their liver, kidneys tests, or if they fail to consume more than 10% of their capsules in weekly monitoring.

Subjects will be randomly assigned to one of two intervention groups (Narangenin capsules) or a control group receiving a placebo. Patient assignment will be conducted using the stratified permuted block randomization method. Patients will be randomly assigned to one of two intervention groups (narangenin capsules) or a control group (placebo) based on their history of diabetes. Each stratum will consist of four cases, with two cases assigned to the placebo group and two cases assigned to the naringenin group. To ensure the blinding of the study, the capsules will be identical in appearance and packaged in the same containers. Each capsule of the intervention group will contain 250 mg of naringenin, while each capsule of the control group will contain 250 mg of starch. The capsules are administered to the patients by the nursing staff, who are unaware of the patient grouping. The supplementation regimen will commence one day following surgery, with participating patients receiving two capsules (equivalent to 500 mg) daily for 14 days. Subsequently, following a 14-day period, the patients will resume the maintenance dose of 250 mg per day until the 90th day post-surgery. During the intervention period, patients will be monitored for regular use of the capsules and any adverse reactions. Patients will be required to attend the hospital's orthopedic clinic on two occasions: 14 days after surgery and three months after surgery. During these visits, fasting blood samples will be taken for biochemical tests. The fusion status of patients will be evaluated by radiography after surgery, 14 days, and three months after surgery. Additionally, functional testing (Oswestry disability index (ODI)) will be performed two weeks and three months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for orthopedic surgery for bone fractures of the lower limbs,
* Ambulatory without assistance for a minimum of two months prior to the fracture.
* Not having undergone amputation of the lower limbs.
* Not suffering from liver cirrhosis.
* Not suffering from advanced kidney failure (blood creatinine higher than 1.4 mg/dL).
* Not having metastatic cancer, any chronic inflammatory diseases, nor taking any drugs that affect bone metabolism, including calcitonin, bisphosphonates, and corticosteroids.

Exclusion Criteria:

* Allergy or intolerant reaction to narangenin capsules
* Any abnormal changes in their liver, kidneys tests,
* Failure to consume more than 10% of their capsules

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-03 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
Circulating inflammatory markers | Baseline, 14 days post-surgery, and 90 days post-surgery.
  Plasma or serun inflammatory merkers including c-reactive protein and pentraxin 3

SECONDARY OUTCOMES:
The rate of bone fusion | Baseline, 14 days post-surgery, and 90 days post-surgery.
Oswestry disability index | Baseline, 14 days post-surgery, and 90 days post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ayatollah Taleghani Educational Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No